CLINICAL TRIAL: NCT01308632
Title: PHASE I-II TRIAL OF METRONOMIC TEMOZOLAMIDE WITH INTERMITTENT INTENSIFICATION AND IRINOTECAN IN PATIENTS WITH RECURRENT GLIOBLASTOMA
Brief Title: Metronomic Temozolamide in Patients With Recurrent Glioblastoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo Español de Investigación en Neurooncología (Other)
Responsible Party: Grupo Español de Investigación en Neurooncología,, GEINO
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GENOM-007
Record Dates: First submitted 2011-01-24; First posted 2011-03-04 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Glioblastoma
Keywords: glioblastoma; temozolamide; radiotherapy; TMZ; irinotecan
MeSH Terms: conditions — Glioblastoma | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temozolamide, irinotecan (Experimental): Phase I trial:
  TMZ will be administered in a fixed schedule as follows:
  TMZ 50 mg/m2/day divided in three daily doses (approx. 17 mg/m2/8 hours) on days 1-7, 9-21, and 23-28.
  100 mg/m2 in a morning single dose on days 8 and 22
  CPT-11 starting dose:
  100 mg/m2 on days 8 and 22, administered 3 to 6 hours after TMZ. (Level 1)
  One cycle = 28 days
  CPT-11 will be escalated in successive cohorts of 3 patients as follows: 115, 130, 145, 160 mg/m2 .
  Interventions: Drug: Temozolamide, irinotecan

INTERVENTIONS:
Drug: Temozolamide, irinotecan — Phase I trial:
  TMZ will be administered in a fixed schedule as follows:
  TMZ 50 mg/m2/day divided in three daily doses (approx. 17 mg/m2/8 hours) on days 1-7, 9-21, and 23-28.
  100 mg/m2 in a morning single dose on days 8 and 22
  CPT-11 starting dose:
  100 mg/m2 on days 8 and 22, administered 3 to 6 hours after TMZ. (Level 1)
  One cycle = 28 days
  CPT-11 will be escalated in successive cohorts of 3 patients as follows: 115, 130, 145, 160 mg/m2 .
  Other Names: CPT-11; Campto; Irinotecan; Temozolamide

SUMMARY:
Indication:

Subjects with glioblastoma at first relapse after surgery, radiotherapy and first-line temozolomide (TMZ).

Objectives:

1. Phase I endpoint:

   - To determine the maximum tolerated dose (MTD) of CPT-11 administered on days 8 and 22 in combination with a fixed, continuous, and metronomic regimen of TMZ, given in 28-day cycles.
2. Phase II endpoints:

Primary endpoint: Progression-free survival at 6 months. Secondary endpoints: Response rate, toxicity profile, overall survival.

Complementary studies:

To assess the effect of treatment on plasma concentration of thrombospondin-1 (TSP1), soluble VEGF receptor 1 (sVEGF-1) and VEGF-A, and their correlation with clinical outcome.

* To assess the correlation between immunohistochemical expression of PTEN and MGMT proteins, and clinical outcomes.

DETAILED DESCRIPTION:
Study Design: Open label, phase I - II trial. Phase I trial: TMZ will be administered in a fixed schedule as follows:

TMZ

* 50 mg/m2/day divided in three daily doses (approx. 17 mg/m2/8 hours) on days 1-7, 9-21, and 23-28.
* 100 mg/m2 in a morning single dose on days 8 and 22

CPT-11 starting dose:

.100 mg/m2 on days 8 and 22, administered 3 to 6 hours after TMZ.(Level 1).One cycle = 28 days. CPT-11 will be escalated in successive cohorts of 3 patients as follows: 115, 130, 145, 160 mg/m2 .

Three patients will be treated at dose level 1. If there is no DLT, 3 new patients will be treated at dose level 2, and so on. If 1 or 2 of the 3 patients initially recruited at each treatment level experience DLT, 3 additional patients will be included at the same level. If DLT is registered in less than 3 of the 6 patients treated at this level, 3 new patients will be included in the next dose level. If 3 or more of the 6 patients experience DLT, the phase I trial will be closed and the previous treatment level will be chosen for the phase II trial. If all 3 initial patients at one level experience DLT, the previous dose level will be used in the phase II trial.

If DLT is found at dose level 1, phase I trial will be re-started at level -2 (70 mg/m2 ) and -1 (85 mg/m2).

Definition of DLT:

* Absolute neutrophil count (ANC) < 500/ μl > 7 days
* Platelet count < 25000/ μl
* A delay in starting a new cycle by > 7 days to allow recovery from toxicity (ANC ≥ 1500/ μl and platelet count ≥ 100000/ μl
* Febrile Neutropenia
* Non-haematological toxicity grade 3-4, except alopecia and nausea/vomiting or diarrhea without adequate prophylaxis or treatment.

Phase II trial: Patients will receive the treatment schedule at the dose level stated in the phase I study. Treatment will be maintained until progression or excessive toxicity.

Patient evaluation: A physical examination, blood count, and basic biochemistry assessment will be performed within 3 weeks before treatment and at each study visit. Tumor recurrence or progression has to be demonstrated by MRI scan performed within 3 weeks before the first treatment course and after every second course of chemotherapy. The assessment of tumor response will be based on criteria defined by Macdonald et al. Study visits will be performed on days 1, 8, 15 and 22 of first and second treatment course, and on days 8 and 22 thereafter, if no significant toxicity has been observed.

Complementary studies: The immunohistochemical expression of PTEN and MGMT will be assessed in paraffin sections of tumor tissue of all patients.

Blood samples for enzyme immunoassay of TSP1, sVEGFR-1 and VEGF-A will be collected within 3 weeks before treatment, after course 1 and every 3 treatment courses thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years old
2. Histological confirmed GB at first relapse, assessed by MRI scan, after surgical resection or biopsy, radiotherapy, and first-line chemotherapy with TMZ. A TMZ treatment duration of at least 3 months is required. Previous chemotherapy with CPT-11 is not allowed.
3. Karnofsky performance status ≥ 70.
4. ANC ≥ 1500/ μl, platelet count ≥ 100000/ μl, haemoglobin > 10 g/dl, serum creatinine and total bilirubin < 1.5 times the upper limit of laboratory normal, transaminases < 3.0 times the upper limit of laboratory normal.
5. Stable or descending corticosteroid dose ≥ 72 hours before baseline MRI and study treatment.
6. Life expectancy greater than 3 months
7. Written informed consent.

Exclusion Criteria:

1. Pregnancy or breastfeeding.
2. Neurological impairment that precludes comprehension or treatment administration
3. Vomiting or other condition that interfere with oral administration of TMZ
4. Previous or concurrent malignancy, excluding basal cell carcinomas or in situ cervical cancer.
5. Concurrent disease that could interfere with treatment
6. Concurrent treatment with enzyme-inducing drugs. Patients under enzyme-inducing anticonvulsants should discontinue treatment at least one week before study treatment and begin a new anti-epileptic treatment with non enzyme-inducing drugs if indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-11; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the treatment (Phase I) | every patient should receive at least one cycle ( 28 days)
  To determine the maximum tolerated dose (MTD) of CPT-11 administered on days 8 and 22 in combination with a fixed, continuous and metronomic regimen of TMZ, given in 28-days cycles to use the Recommended Dose in phase II
Progression-free survival (Phase II) | Since the initial of the treatment until the patient progression
  The time the patient is not in progression, since the beginning of the treatment

SECONDARY OUTCOMES:
Assess the toxicity of the treatment | the patients will be followed until disease progression
  Toxicity Profile (in phase II)
Progression-free survival at 6 months | 6 months since the pacient is included in the trial
  Progression-free survival at 6 months (Phase I)
overall survival | the patients will be followed until death

CONTACTS AND LOCATIONS:
Overall Officials: Reynés Gaspar, Dr, Principal Investigator — Hospital Universitario La Fe de Valencia